CLINICAL TRIAL: NCT02129556
Title: A Phase Ib/II Trial Evaluating the Efficacy of MK-3475 and Trastuzumab in Patients With Trastuzumab-resistant, HER2-positive Metastatic Breast Cancers
Brief Title: Anti-PD-1 Monoclonal Antibody in Advanced, Trastuzumab-resistant, HER2-positive Breast Cancer
Acronym: PANACEA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 45-13 / BIG 4-13; 2013-004770-10 (EudraCT Number)
Record Dates: First submitted 2014-04-24; First posted 2014-05-02 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic; Breast; trastuzumab-resistant; PD-L1 expressing; HER2-positive
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MK-3475 with trastuzumab (single arm) (Experimental): Phase Ib: MK-3475 at dose of 2 mg/kg or 10 mg/kg (i.v.), or a fall-back dose of 1 mg/kg, together with trastuzumab 6mg/kg by (i.v.) once every 3 weeks.
  Phase II: MK-3475 at a flat dose of 200mg (i.v.) together with trastuzumab 6mg/kg (i.v.) once every 3 weeks until progression, lack of tolerability, or 24 months of treatment.
  A dose of 8mg/kg trastuzumab will be used in cycle 1 if prior treatment with trastuzumab was stopped more than 3 months before.
  Interventions: Drug: MK-3475

INTERVENTIONS:
Drug: MK-3475 — The phase Ib trial will determine the recommended dose from three MK-3475 dose levels: 1mg/kg, 2 mg/kg or 10 mg/kg.
  Other Names: Pembrolizumab

SUMMARY:
Panacea is a phase Ib/II trial evaluating the efficacy of MK-3475 and trastuzumab in patients with trastuzumab-resistant, HER2- positive metastatic breast cancers

DETAILED DESCRIPTION:
A significant amount of preclinical and correlative clinical data suggest that HER2-positive breast cancer could be amenable to immune¬therapeutic approaches. The presence of HER2-overexpression in breast cancers is associated with higher levels of proliferation, high histologic grade and higher levels of tumor infiltrating lymphocytes (TILs) compared with HER2-negative tumors. The investigators therefore hypothesize that for HER2-positive tumors, avoidance of destruction by the host immune system must be an important mechanism contributing to tumor growth and progression.

The term "immune evasion" refers to the ability of the tumor to suppress and change host anti-tumor immune reactions. The programmed cell death 1 (PD-1) pathway represents a major immune control switch which may be engaged by tumor cells to overcome active T-cell immune surveillance. The ligands for PD-1 (PD-L1 and PD-L2) are constitutively expressed or can be induced in various tumors. High expression of PD-L1 on tumor cells (and to a lesser extent of PD-L2) has been found to correlate with poor prognosis and survival in various other solid tumor types. Furthermore, PD-1 has been suggested to regulate tumor-specific T-cell expansion in patients with malignant melanoma. These observations suggest that the PD-1/PD-L1 pathway plays a critical role in the tumor immune evasion and could be considered an attractive target for therapeutic intervention in several solid organ types.

MK-3475 (previously known as SCH 900475) is a potent and highly-selective humanized mAb of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. MK-3475 strongly enhances T lymphocyte immune responses in cultured blood cells from healthy human donors, cancer patients, and primatesMK-3475 also modulates the level of interleukin-2 (IL-2), tumor necrosis factor alpha (TNFα), interferon gamma (IFNγ), and other cytokines.

The investigators therefore propose to evaluate if the addition of an immunotherapy can reverse trastuzumab resistance and improve clinical outcomes in HER2-positive disease. In this study the investigators will determine if a monoclonal antibody targeted against PD-1, a T cell negative regulator, can reverse trastuzumab resistance in patients previously progressing on trastuzumab.

ELIGIBILITY:
Inclusion criteria for screening:

* Female gender
* Age ≥ 18 years
* Histologically confirmed breast adenocarcinoma that is unresectable loco-regional, or metastatic.
* Locally confirmed HER2-positivity (immunohistochemistry score 3+) or ERBB2-amplification (Ratio ERBB2/centromeres ≥2.0 or mean gene copy number ≥ 6) of primary tumor or of biopsy from metastatic or unresectable loco-regional lesion.
* Trastuzumab resistant disease, defined by:

  * progression of disease while on-treatment with trastuzumab
  * recurrence while on adjuvant trastuzumab or within 12 months of completing adjuvant trastuzumab
  * Any number of prior lines of anti-HER2 therapy acceptable. Patients for whom the treatment with the current first-line combination of trastuzumab, pertuzumab and taxanes is not an option can be considered for enrollment
* If a patient has received a subsequent anti-HER2 therapy, she must also have progressed on the subsequent therapy.
* Presence of at least one measurable lesion (RECIST 1.1)
* LVEF ≥50%
* Patient agrees to submit an FFPE tumor biopsy for central confirmation of HER2 positivity and central assessment of PD-L1 status.
* Written Informed Consent (IC) for screening procedures and trial participation must be signed and dated by the patient and the Investigator prior to screening.
* Written consent to biological material submission, indicating the patient has been informed of and agrees to tissue and blood material use, transfer and handling, must be signed and dated by the patient and the investigator prior to any procedures specific for this trial, including consent to translational research on FFPE and fresh frozen tumor biopsies in case the patient is enrolled into the trial.
* The patient has been informed of and agrees to data transfer and handling, in accordance with national data protection guidelines.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Life expectancy >3 months.
* Hematopoietic status:

  * Absolute neutrophil count ≥ 1.5 × 109/L,
  * Platelet count ≥ 100 × 109/L,
  * Hemoglobin ≥ 9 g/dL
* Hepatic status:

  * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN). In the case of known Gilbert's syndrome, a higher serum total bilirubin (< 2 × ULN) is allowed.
  * AST and ALT ≤ 2.5 × ULN; if the patient has liver metastases, ALT and AST must be ≤ 5 × ULN.
* Renal status:

  * Creatinine ≤ 1.5 ×ULN or creatinine clearance > 60 ml/min
  * Proteinuria <1 g/day
* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or PTT (partial thromboplastin time) is within therapeutic range of intended use of anticoagulant.

Inclusion criteria for enrollment:

All inclusion criteria for screening, plus:

* Central lab confirmation on a metastatic biopsy (or biopsy from unresectable loco-regional disease) of:

  * HER2-positivity (immunohistochemistry score 3+) or ERBB2- amplification (Ratio ERBB2/centromeres ≥2.0 or mean gene copy number ≥ 6),
  * Presence of PD-L1 expression assessed by IHC (during the phase II portion of the trial a parallel, secondary cohort of 15 patients with PD-L1 negative disease will be enrolled)
* Patient agrees to submit tumor tissue for translational research:

  * tissue biopsy from unresectable loco-regional or metastatic disease obtained ≤1 year prior to enrollment or new tissue material from a recently obtained surgical or diagnostic biopsy. For patients who have presented with stage 4 disease de novo, a biopsy taken from the presumed primary breast lesion is acceptable (provided this was taken ≤1 year prior to enrollment).
  * if available: FFPE tumor block from primary surgery or diagnostic biopsy.
  * if available: pre-treatment fresh frozen tumor biopsy.
  * if feasible: FFPE tumor block from post-treatment biopsy will be taken at time of disease progression or end of all treatment if ended prior to progression. This re-biopsy is strongly advised.
  * if feasible: fresh frozen tumor biopsy from post-treatment biopsy will be taken at time of disease progression or end of all treatment if ended prior to progression.
* Patient agrees to submit baseline (pre-treatment) blood and serial plasma for translational research
* For patient of childbearing potential, negative serum pregnancy test. Pregnancy test has to be repeated within 72h before treatment start.
* All anti-cancer treatment including endocrine therapy, with the exception of trastuzumab, must stop 3 weeks prior to first dose of trial treatment.

Exclusion criteria for screening:

* Prior therapy with other anti-PD-1, anti- PD-L1, L2 or anti-CTLA4 therapy.
* No FFPE material to centrally assess HER2-positivity and PD-L1 expression.
* Known Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), or positive for Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA [qualitative]).
* Interstitial lung disease
* History of or active pneumonitis requiring treatment with steroids
* Active central nervous system metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth (patients with history of CNS metastases or spinal cord compression are eligible if they are clinically and radiologically stable for at least 4 weeks before first dose of investigational product and have not required high-dose steroid treatment in the last 4 weeks).
* Leptomeningeal disease
* History of clinically significant or uncontrolled cardiac disease, including congestive heart failure (New York Heart Association functional classification ≥3), angina, myocardial infarction or ventricular arrhythmia.
* Previous severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Active infection requiring systemic therapy.
* Chronic systemic therapy with immunosuppressive agents including cortico¬steroids.
* Concurrent disease or condition that would make the patient inappropriate for trial participation or any serious medical disorder that would interfere with the patient's safety.
* Known history of uncontrolled hypertension (≥ 180/110), unstable diabetes mellitus, dyspnea at rest, or chronic therapy with oxygen.
* Dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of Informed Consent.
* Treatment with an investigational agent in the 4 weeks before enrollment.
* Active autoimmune disease or a documented history of autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the trial. Patients with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the trial.
* Chemotherapy, radioactive therapy, and/or biological cancer therapy within 3 weeks prior to the first trial dose and has not recovered to CTCAE v.4 grade 1 or better from adverse events.
* Pregnant or lactating women; lactation has to stop before enrollment.
* The patient of childbearing potential who is unwilling to use highly effective contraception during treatment and up to 7 months after stop of trial treatment. Acceptable methods are intrauterine devices (without hormones), bilateral tubal occlusion, vasectomized partner or total abstinence. Oral, injectable, or implant hormonal contraceptives are not allowed.
* Unresolved or unstable, serious adverse events from prior administration of another investigational drug.
* Active or uncontrolled infection CTCAE v.4 grade 2 or higher.
* Live vaccines within 30 days prior to the first dose of trial therapy and during trial treatment.

Exclusion criteria for enrollment:

* All exclusion criteria for screening apply for enrollment as well. Excluded are especially patients who have received any of the treatments below:
* Live vaccines within 30 days prior to the first dose of trial therapy and during trial treatment.
* History of CNS metastases or spinal cord compression if they have not been clinically stable for at least 4 weeks before first dose of investigational product and require high-dose steroid treatment.
* Treatment with an investigational agent in the 4 weeks before enrollment.
* Patient has not recovered to CTCAE v.4 grade 1 or better from adverse events of prior therapy, except alopecia grade 2.
* Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), or positive for Hepatitis B or Hepatitis C.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-12; Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherene Loi, MD, Study Chair — Department of Medical Oncology,Peter MacCallum Cancer Centre,East Melbourne, Victoria, Australia; Fabrice André, Prof., Study Chair — Department of Medical Oncology Institut Gustave Roussy,Villejuif,France
Locations (11):
- Australia (2):
  - Peter MacCallum Cancer Centre, East Melbourne
  - Westmead Hospital, Westmead
- Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - Jules Bordet Institute, Brussels
  - CHU Sart Tilman, Liège
- France (4):
  - Institut de Cacérologie de l'OUEST, Angers
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - Istituto Europeo di Oncologia, Milan
  - Azienda USL4 Prato, Prato

REFERENCES:
- [Background] Slamon DJ, Leyland-Jones B, Shak S, Fuchs H, Paton V, Bajamonde A, Fleming T, Eiermann W, Wolter J, Pegram M, Baselga J, Norton L. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med. 2001 Mar 15;344(11):783-92. doi: 10.1056/NEJM200103153441101. PMID 11248153
- [Background] Hurvitz SA, Betting DJ, Stern HM, Quinaux E, Stinson J, Seshagiri S, Zhao Y, Buyse M, Mackey J, Driga A, Damaraju S, Sliwkowski MX, Robert NJ, Valero V, Crown J, Falkson C, Brufsky A, Pienkowski T, Eiermann W, Martin M, Bee V, Marathe O, Slamon DJ, Timmerman JM. Analysis of Fcgamma receptor IIIa and IIa polymorphisms: lack of correlation with outcome in trastuzumab-treated breast cancer patients. Clin Cancer Res. 2012 Jun 15;18(12):3478-86. doi: 10.1158/1078-0432.CCR-11-2294. Epub 2012 Apr 13. PMID 22504044
- [Background] Denkert C, Loibl S, Noske A, Roller M, Muller BM, Komor M, Budczies J, Darb-Esfahani S, Kronenwett R, Hanusch C, von Torne C, Weichert W, Engels K, Solbach C, Schrader I, Dietel M, von Minckwitz G. Tumor-associated lymphocytes as an independent predictor of response to neoadjuvant chemotherapy in breast cancer. J Clin Oncol. 2010 Jan 1;28(1):105-13. doi: 10.1200/JCO.2009.23.7370. Epub 2009 Nov 16. PMID 19917869
- [Background] Loi S, Sirtaine N, Piette F, Salgado R, Viale G, Van Eenoo F, Rouas G, Francis P, Crown JP, Hitre E, de Azambuja E, Quinaux E, Di Leo A, Michiels S, Piccart MJ, Sotiriou C. Prognostic and predictive value of tumor-infiltrating lymphocytes in a phase III randomized adjuvant breast cancer trial in node-positive breast cancer comparing the addition of docetaxel to doxorubicin with doxorubicin-based chemotherapy: BIG 02-98. J Clin Oncol. 2013 Mar 1;31(7):860-7. doi: 10.1200/JCO.2011.41.0902. Epub 2013 Jan 22. PMID 23341518
- [Derived] Loi S, Giobbie-Hurder A, Gombos A, Bachelot T, Hui R, Curigliano G, Campone M, Biganzoli L, Bonnefoi H, Jerusalem G, Bartsch R, Rabaglio-Poretti M, Kammler R, Maibach R, Smyth MJ, Di Leo A, Colleoni M, Viale G, Regan MM, Andre F; International Breast Cancer Study Group and the Breast International Group. Pembrolizumab plus trastuzumab in trastuzumab-resistant, advanced, HER2-positive breast cancer (PANACEA): a single-arm, multicentre, phase 1b-2 trial. Lancet Oncol. 2019 Mar;20(3):371-382. doi: 10.1016/S1470-2045(18)30812-X. Epub 2019 Feb 11. PMID 30765258

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase Ib 2 mg/kg; Phase Ib 10 mg/kg: HER2-positive, PD-L1 expressing, unresectable loco-regional or metastatic breast carcinoma that progressed on prior trastuzumab-based therapy. In the Phase Ib portion of the trial, two weight-based doses of MK-3475 were specified in the dose escalation (2 mg/kg and 10 mg/kg).
- Phase II PD-L1+: HER2-positive, PD-L1 expressing, unresectable loco-regional or metastatic breast carcinoma that progressed on prior trastuzumab-based therapy. The Phase II portion of the trial used a flat dose of 200 mg of MK-3475 based on emerging data from the sponsor.
- Phase II PD-L1-: HER2-positive, PD-L1 negative, unresectable loco-regional or metastatic breast carcinoma that progressed on prior trastuzumab-based therapy. The Phase II portion of the trial used a flat dose of 200 mg of MK-3475 based on emerging data from the sponsor.
Period: Overall Study
Arm/Group | Phase Ib 2 mg/kg | Phase Ib 10 mg/kg | Phase II PD-L1+ | Phase II PD-L1-
Started | 3 | 3 | 40 | 12
Completed | 3 | 3 | 37 | 12
Not Completed | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase Ib; Phase II PD-L1+: HER2-positive, PD-L1 expressing, unresectable loco-regional or metastatic breast carcinoma that progressed on prior trastuzumab-based therapy
- Phase II PD-L1-: HER2-positive, PD-L1 negative, unresectable loco-regional or metastatic breast carcinoma that progressed on prior trastuzumab-based therapy
- Total: Total of all reporting groups
Arm/Group | Phase Ib | Phase II PD-L1+ | Phase II PD-L1- | Total
Number analyzed (Participants) | 6 | 40 | 12 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9.5) | 51.2 (10.4) | 54.5 (5.2) | 51.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 40 | 12 | 58
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 30 | 8 | 42
  Asian | 0 | 2 | 1 | 3
  Other | 0 | 1 | 0 | 1
  Missing | 2 | 7 | 3 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 0 | 0 | 1 | 1
  Belgium | 0 | 6 | 3 | 9
  Italy | 0 | 6 | 1 | 7
  Australia | 4 | 13 | 4 | 21
  France | 2 | 15 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Dose-Limiting Toxicity (DLT) of MK-3475 in Combination With Trastuzumab
Description: Determination of dose-limiting toxicity (DLT) which is defined as an adverse event or abnormal laboratory value assessed as suspected to be trial treatment related (possible, probable or definite) and unrelated to disease or disease progression. Toxicities and lab values will be graded according to the NCI CTCAE (v4.0).
  1. Any grade-3 or greater non-hematological adverse event lasting at least one week;
  2. Any grade-4 hematological toxicity; or,
  3. Any adverse event resulting in a delay starting cycle 2 of more than 14 days.
Time Frame: Within the first 21 days
Population: Patients enrolled during phase Ib portion, a patient receiving one or more doses of MK-3475 and trastuzumab is considered evaluable.
Measure: Count of Participants; unit: Participants
Groups:
- Phase Ib 2 mg/kg; Phase Ib 10 mg/kg: HER2-positive, PD-L1 expressing, unresectable loco-regional or metastatic breast carcinoma that progressed on prior trastuzumab-based therapy
Arm/Group | Phase Ib 2 mg/kg | Phase Ib 10 mg/kg
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

2. Primary Outcome: Objective Response Rate (ORR)
Description: Confirmed CR or PR as best overall response. At the time of each restaging, patients will be classified as achieving complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or non-evaluable for response according to RECIST (Version 1.1) criteria.
Time Frame: Clinical and radiological tumor assessment will be performed by CT scan or MRI at baseline, at weeks 12, 18 and 24, then every 12 weeks until progression, or 24 weeks after stop of treatment if before progression.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Groups:
- Phase Ib: HER2-positive, PD-L1 expressing, unresectable loco-regional or metastatic breast carcinoma that progressed on prior trastuzumab-based therapy. All 6 patients in Phase Ib were combined when reporting clinical measures for secondary outcomes and adverse events, for stronger response rates.
Arm/Group | Phase Ib | Phase II PD-L1+ | Phase II PD-L1-
Number analyzed (Participants) | 6 | 40 | 12
proportion of participants | 0.17 [0.01 to 0.58] | 0.15 [0.07 to 0.29] | 0.00 [0.00 to 0.18]

3. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response (DoR) is defined among patients with objective response (confirmed CR or PR as best overall response) as the interval between dates of first documentation of objective response and first documentation of progressive disease. In the absence of documented progressive disease, follow-up will be censored at date of last disease assessment.
Time Frame: From date of first documentation of objective response until first documentation of progressive disease, up to 24 weeks after stop of treatment (=30 months)
Population: Patients who achieved objective response
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase Ib | Phase II PD-L1+ | Phase II PD-L1-
Number analyzed (Participants) | 1 | 6 | 0
months | 23.1 | 3.5 [2.7 to 999999] |

4. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) defined as the interval between the dates of the start of trial treatment and first documentation of progressive disease. In the absence of documented progressive disease, follow-up will be censored at date of last disease assessment
Time Frame: From the first trial treatment until first documentation of progressive disease up to 24 weeks after stop of treatment (=30 months)
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase Ib | Phase II PD-L1+ | Phase II PD-L1-
Number analyzed (Participants) | 6 | 40 | 12
months | 2.5 [1.1 to 2.7] | 2.7 [2.6 to 4.9] | 2.5 [1.4 to 999999]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: The proportion of patients with best confirmed RECIST response of CR, PR, or duration of SD of at least 24 weeks (measured from first dose of trial treatment).
Time Frame: From the start of trial treatment until confirmed CR, PR, or SD lasting for 24 weeks or longer
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Phase Ib | Phase II PD-L1+ | Phase II PD-L1-
Number analyzed (Participants) | 6 | 40 | 12
proportion of participants | 0.17 [0.01 to 0.58] | 0.25 [0.14 to 0.39] | 0.00 [0.00 to 0.18]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: The interval between the dates of the first dose of trial treatment until first documentation of disease progression or death, whichever occurs first. Patients with new non-breast cancer malignancy must continue to be followed for progression of the original breast cancer. For patients without progression, follow-up is censored at the date of last disease assessment without progression, unless death occurs within 12 weeks following the date last known progression-free, in which case the death will be counted as a PFS event.
Time Frame: From the date of first treatment dose until documented disease progression or death from any cause. whichever occur first, assessed up to 30 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase Ib | Phase II PD-L1+ | Phase II PD-L1-
Number analyzed (Participants) | 6 | 40 | 12
months | 2.5 [1.1 to 2.7] | 2.7 [2.6 to 4.0] | 2.5 [1.4 to 2.7]

7. Secondary Outcome: Overall Survival (OS) at 12 Months
Description: OS is defined as the time from the first dose of trial treatment to death from any cause. For patients who are lost to follow-up or who have no documentation of death at the time of final analysis, follow-up is censored at the date of last assessment of vital status. OS at 12 months by Kaplan-Meier estimates.
Time Frame: Time from start of trial treatment to death from any cause, assessed up to 30 months
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Phase Ib | Phase II PD-L1+ | Phase II PD-L1-
Number analyzed (Participants) | 6 | 40 | 12
proportion of participants | 0.67 [0.27 to .88] | .65 [.50 to .76] | .12 [.01 to .36]

ADVERSE EVENTS:
Time Frame: From the date of signature of informed consent until 30 days after all treatment discontinuation, regardless of whether it was considered related to a medication. AEs were to be reported at the end of every treatment cycle, at the End-of-Treatment visit, and up to 30 days after cessation of trial treatment. Serious adverse event and pregnancy data were to be collected for 90 days following the end of treatment.
Description: Any grade of any observed AE was to be reported on the AE form. There were no specifications of targeted AEs. Symptoms of the targeted cancer were not to be reported as AEs. AEs were categorized and graded according to CTCAE V4.
Groups:
- Phase Ib: HER2-positive, PD-L1 expressing, unresectable loco-regional or metastatic breast carcinoma that progressed on prior trastuzumab-based therapy. All 6 patients in Phase I were combined when reporting clinical measures for secondary outcomes adverse events for stronger response rates.
- Phase II (PD-L1+ and PD-L1-): HER2-positive, PD-L1 expressing or PD-L1 negative, unresectable loco-regional or metastatic breast carcinoma that progressed on prior trastuzumab-based therapy. For adverse events, Phase II cohorts were combined since PD-L1 status does not affect toxicity.
Arm/Group | Phase Ib | Phase II (PD-L1+ and PD-L1-)
All-Cause Mortality (participants affected / at risk) | 4/6 | 25/52
Serious Adverse Events (participants affected / at risk) | 4/6 | 25/52
Other Adverse Events (participants affected / at risk) | 6/6 | 50/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib (N=6) | Phase II (PD-L1+ and PD-L1-) (N=52)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Takotsubo cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CNS metastases (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Disease progression (Reproductive system and breast disorders) | 2 (2) | 6 (6)
Death (General disorders) | 2 (2) | 9 (9)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Breast infection (Reproductive system and breast disorders) | 0 | 1 (1)
Bile duct dilatation (Hepatobiliary disorders) | 0 | 1 (1)
Catheter-related infection (Infections and infestations) | 0 | 1 (1)
Sepsis (Infections and infestations) | 0 | 1 (1)
Plural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 (3)
Intracranial hypertension (Vascular disorders) | 0 | 1 (1)
Cognitive disturbance (Psychiatric disorders) | 0 | 1 (1)
Acute renal impairment (Renal and urinary disorders) | 0 | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 | 2 (2)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 (3)
Lambert-Eaton syndrome (Immune system disorders) | 0 | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 | 1 (1)
GGT increased (Investigations) | 0 | 1 (1)
Paresthesia (Nervous system disorders) | 0 | 1 (1)
Neurological paresis (Nervous system disorders) | 0 | 1 (1)
Aphasia (Nervous system disorders) | 0 | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 (1)
Autoimmune hepatitis (Immune system disorders) | 0 | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib (N=6) | Phase II (PD-L1+ and PD-L1-) (N=52)
Anemia (Blood and lymphatic system disorders) | 4 (6) | 8 (8)
Fever (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Reactive thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Takotsubo cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (3) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1)
Visual field defect left lower quadrants (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Abdominal pain, intermittent (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 2 (5) | 9 (11)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (2) | 11 (14)
Nausea with weight loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue mycosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4)
Anemia (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Diaphoresis (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 4 (4)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 16 (23)
Fever (General disorders) | 1 (1) | 3 (5)
Flu-like symptoms (General disorders) | 0 (0) | 5 (5)
Hoarseness (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Left breast tumour bleeding (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (4)
Pain (General disorders) | 0 (0) | 6 (10)
Bile duct dilatation (Hepatobiliary disorders) | 0 (0) | 1 (2)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 3 (3)
Catheter-related infection (Infections and infestations) | 1 (1) | 1 (1)
Dental (Infections and infestations) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (4)
Rhinitis infective (Infections and infestations) | 0 (0) | 3 (4)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (4) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (3)
Yeasts in the stool (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (3)
Drug induced liver injury (Investigations) | 0 (0) | 1 (1)
Ggt increased (Investigations) | 0 (0) | 5 (11)
Hypercalcemia (Investigations) | 0 (0) | 1 (1)
Leucocyte count decreased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 3 (6)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Serum amylase increased (Investigations) | 0 (0) | 3 (3)
Weight loss (Investigations) | 0 (0) | 4 (4)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Aphonia (Nervous system disorders) | 0 (0) | 1 (2)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 8 (15)
Loss of hand motor traction (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Static cerebellar syndrom (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Acute renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 11 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis: seasonal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Cutaneous rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (7)
Cutaneous toxicity on legs and arms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erysipelas (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
Rash - face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Redness ankle and feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 6 (12)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Intracranial hypertension (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema right leg (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-04-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT02129556/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT02129556/SAP_001.pdf